CLINICAL TRIAL: NCT01311154
Title: Impact of Specific Antibiotic Therapies on the Prevalence of Human Host Resistant Bacteria - WP5
Brief Title: Impact of Specific Antibiotic Therapies on the Prevalence of Human Host Resistant Bacteria
Acronym: SATURN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: European Union (Other)
Responsible Party: yehuda carmeli, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-0425-10-TLV
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Focus of Study: Carriers of Resistant Enterobacteriaceae.
Keywords: carriers; resistant Enterobacteriaceae; AMR; antibiotic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The proposed study is distinctive in studying known carriers of resistant Enterobacteriaceae. It examines both phenotypic and genotypic expansion in the AMR bacterial population as a function of antibiotic treatment, and examines the effect of antibiotics on the dissemination of resistance genes from species to species. It will examine CRE, important emerging pathogens, which are a significant threat to public health, but yet not well studied. The proposed study will use an interdisciplinary approach, combining PK/PD, phenotypic, and genetic data to understand the effect of antibiotics on the likelihood of spread of AMR. Most previous studies have focused on the effect of antibiotic agents on clinical detection, infection or acquisition of AMR among non-carriers67,68. Other studies have looked at the effects on colonisation-resistance mostly among healthy volunteers69. Very few studies have examined the effects of various antibiotic agents on carriers of ARB and those focused primarily on vancomycin resistant enterococci (VRE)70. No similar studies have been conducted with regard to ESBL or to CRE. Correlation with clinical factors and environmental contamination has not been determined in previously published studies. The proposed study also extends the analysis to the effect of antibiotic treatment on dissemination of resistance genes which may be of great importance as these events may lead to emergence of new AMR strains and species. The proposed study not only examines the effects of various antibiotic agents and classes, but also the effects of duration of treatment and PK/PD indices on amplification of ARB. The study will also examine the effect of antibiotics on the epidemicity and fitness of colonising strains

DETAILED DESCRIPTION:
We will conduct an observational longitudinal prospective study in 3 hospitals in units with high prevalence of resistant organisms. Consenting patients will be screened for carriage of AMR organisms at admission, and those found to be carriers of the target ARB will be included in the longitudinal study. To improve the yield of screening we may use risk stratification based on risk factors identified at each center. Patients included in the longitudinal study will be asked to provide serial stool samples every 2-3 days during hospitalisation (rectal swab will be allowed as replacement for stool specimen, after developing appropriate methodology to correlate between stool samples and rectal swabs).

These samples will be analysed using quantitative cultures for the number of resistant organisms, and samples will be subject to quantitative real time PCR to quantify resistant genes (CTX-M, TEM, SHV, KPC, VIM as required). In parallel, environmental contamination will be examined and quantified using similar methods. Data will be collected daily regarding antibiotic treatment, other medications, clinical parameters, bowel movements and presence of diarrhoea, and various PK/PD indices. The target antibiotic for this study include commonly use agents in the hospital setting including quinolones, cephalosporins, piperacillin/tazobactam, ertapenem, imipenem, doripenem, metronidazole, clindamycin and aminoglycosides. The duration, the sequential order of treatment and PK/PD indices will be examined. The effects of surgical antibiotic prophylaxis will be examined as an important end point. The effects of the target antibiotic agents/classes on selection, enrichment, and spread of the target AMR organisms. Analyses will be conducted to compare: 1. the effects of various antibiotics 2. the effect of duration of therapy 3. the durability of the effect (posttreatment). 4. The effects of PK/PD indices.

Secondary analysis will examine the risk of developing infections as function of various factors including time and load of carriage of resistant organisms and of exposure to antibiotics will be performed. Correlation with clinical isolates will be performed including typing, gene and plasmid analyses to determine correlation between colonising and infecting strains. Experiment simulating patient contact will be conducted to examine contamination of hands, gloves and gowns after contact in order to correlate between environmental contamination and contamination of healthcare workers. Additional work will be conducted on profiling bacterial communities by DNA fingerprinting techniques using length hetrogeneity (LH-PCR) and automated ribososmal internal spacer analysis (ARISA) on a sample of the patients studied.

ELIGIBILITY:
Inclusion Criteria:

known carriers of resistant Enterobacteriaceae

Exclusion Criteria:

no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: known carriers of resistant Enterobacteriaceae
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-02 (Estimated); Study Completion 2015-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Tasmc, Tel Aviv, Israel